CLINICAL TRIAL: NCT06427616
Title: Effects of Short Duration Moderate Intensity Soleus Pushups Versus Sustained Soleus Pushups on Blood Glucose Level Among Young Population
Brief Title: Moderate Intensity Soleus Pushups Versus Sustained Soleus Pushups on Blood Glucose Level Among Young Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3547 Sara Noor
Record Dates: First submitted 2024-05-06; First posted 2024-05-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Duration Moderate Intensity Soleus Push-ups (Group A) (Experimental): Moderate intensity involving weighted soleus push-ups is performed till patient start to fatigue
  Interventions: Behavioral: Short Duration Moderate Intensity Soleus Push-ups
- Sustained Soleus Push-ups (Group B) (Experimental): Sustained soleus push-ups will be performed for up to 270 min.
  Interventions: Behavioral: Sustained Soleus Push-ups

INTERVENTIONS:
Behavioral: Short Duration Moderate Intensity Soleus Push-ups — participants performed moderate intensity soleus push-ups with ankle weights, calculated as 30-40% of individuals 1RM of soleus muscle's strength. The single set of MSPU was performed 15 minutes after the meal for time till the point where the muscle started to fatigue. The participants were in sitting position with legs positioned at 90 degree angle relative to floor and feet flat on ground performed continuous planter flexion against the ankle weight. Three sets of MSPU was performed at every 15 and Session lasted in 60 minutes.
  Other Names: Group A
  Arms: Short Duration Moderate Intensity Soleus Push-ups (Group A)
Behavioral: Sustained Soleus Push-ups — Participants will start soleus push-ups in sitting. To do so, the participants will be in a seated position, the legs will be at 90 degrees to the floor, and feet will be placed flat on the ground. Participants will then move their heels up and down continuously for.
  Sustained soleus push-ups will be performed with light intensity for up to 270 mins.
  No external resistance will be added. Participants will be provided with a maximum of 4 min break time after every 90 mins intervention. In the meantime, their blood sample will be collected
  Other Names: Group B
  Arms: Sustained Soleus Push-ups (Group B)

SUMMARY:
To determine that the short duration moderate intensity soleus push-ups will have a better effect on blood glucose level as compared to sustained soleus push-ups.

DETAILED DESCRIPTION:
The soleus muscle is a slow oxidative muscle which possesses molecular machinery necessary for regulating blood borne substrates. It has the ability to increase the local oxidative metabolism for a long period of time without experiencing fatigue. The uniqueness lies in this muscle because of its inability to store glycogen and derives its energy directly from the glucose present in the bloodstream. This in turn helps in lowering the blood sugar by using the excess blood glucose as its primary source of fuel. The soleus muscle also stands out because of its high composition of slow oxidative fibers, around 88% of the fibers are slow twitch fibers, making it the only muscle in human body containing greater proportion of slow twitch fiber.

A specific exercise called soleus push-ups (SPU) can have a huge impact on boosting metabolism and regulating blood glucose level better than the total body muscle exercises, intermittent fasting, weight loss etc. According to the previous study it showed a significant effect on the overall blood chemistry when performed for 270 mins.

So,the purpose of this study will be to find the comparison of acute effects of sustained soleus push-ups with moderate resisted soleus push-ups on blood sugar level. To find whether moderate resisted soleus push-ups will give same or better results in short period of time.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* Gender: both male and female.
* Healthy young adults.
* BMI: healthy weight.

Exclusion Criteria:

* Patient with cardiac issues.
* Any neurological issues.
* Knee injuries.
* Patient with any lower limb injuries.
* DVT and lower amputation.
* Any known diabetic patient.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Sugar Level | Baseline to 6 hours
  The primary outcome measure will be the change in blood sugar level, measured before and after the intervention period. This will provide insight into the direct impact of short duration moderate intensity soleus push-ups vs sustained soleus push-ups on blood sugar levels among young individuals.

OTHER OUTCOMES:
Perception, acceptability and feasibility of participants to measure the Adherence | Baseline to 6 hours
  Adherence to the prescribed exercise will be monitored throughout the intervention period to assess compliance and determine if there are any differences in adherence between the two exercise groups.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No